CLINICAL TRIAL: NCT07318220
Title: Optimizing Cancer Support Services Usage in Patients With Head and Neck Cancer During the Prehabilitation Period
Brief Title: Prehabilitation Protocol for Head and Neck Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Akina Natori, Research Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20230516
Record Dates: First submitted 2025-12-22; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aim 2: Prehabilitation Prescription Protocol Group (Experimental): Participants in this group will be referred to a prehabilitation prescription protocol of nutritional counseling and exercise for HNC patients. Participants will attend for nutritional counseling and exercise sessions for the duration of their radiation therapy (RT) or chemoradiation therapy (CRT) for HNC. The duration of these sessions depends on the participant's treatment plan and the timing of enrollment.
  Participants will also have three in-person assessments during the study period during the following timepoints (T), to assess feasibility and acceptability of the prehabilitation prescription protocol: Baseline (T1), at the completion of RT/CRT (T2), and 8 weeks after the completion of RT/CRT and the exit survey (T3).
  Total participation duration is up to 18 weeks.
  Interventions: Behavioral: Referral to Oncology Nutritional Counseling and Exercise Program

INTERVENTIONS:
Behavioral: Referral to Oncology Nutritional Counseling and Exercise Program — Participants will be referred by their healthcare provider to an oncology nutritional counseling and exercise program administered standard of care by the Cancer Support Service at the Sylvester Comprehensive Cancer Center. Participants will be scheduled to the predetermined frequency and length of visits with oncology dietitians and exercise physiologists per the prehabilitation prescription protocol developed during the pre-implementation period.

SUMMARY:
The purpose of this research is to help researchers understand the barriers, supports, and preferences for prehabilitation. Prehabilitation in this study means head and neck cancer patients will receive nutritional counseling sessions and attend exercise programs before and during radiotherapy/chemoradiotherapy treatment.

ELIGIBILITY:
Aim 2 Inclusion Criteria: Implement prehabilitation prescription protocol and evaluate the feasibility and acceptability of the prehabilitation prescription protocol in a sample of HNC patients.

1. Age 18 to 80 years old
2. Patients with a diagnosis of non-metastatic squamous cell carcinoma originating in the head and neck (oral cavity, oropharynx, hypopharynx, larynx, and nasopharynx).
3. Patients with a plan for curative radiation therapy (RT) / chemoradiation therapy (CRT) at SCCC* - *Patients who underwent surgery for the HNC are still eligible.
4. Clearance for exercise by the medical team.
5. Patients who do not have their first treatment scheduled within 3 weeks at the time of recruitment.
6. An English or Spanish speaker.

Aim 2 Exclusion Criteria:

1. A patient with a metastatic cancer.
2. A patient who cannot complete the baseline assessment and/or start prehabilitation by the initiation of RT/CRT.
3. Any contraindication for diet change or exercising as determined by a physician.
4. Engaging in >150 minutes of moderate to vigorous physical activity on average per week for the prior month.
5. A patient who is not an English or Spanish speaker.
6. History of dementia or major psychiatric disease which would interfere with study.
7. History of recent (≤1 yr) stroke, myocardial infarction, or congestive heart failure
8. Eastern Cooperative Oncology Group (ECOG) equal to or higher than 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Aim 2: Feasibility of Participant Engagement in Prehabilitation Prescription Program | Up to 18 Weeks
  Feasibility will be measured as the percentage of participants that agree to participate in the prehabilitation prescription protocol. Criterion for success: At least (≥) 50% of all eligible participants agree to participate in the prehabilitation prescription protocol.
Aim 2: Feasibility of Participant Attendance to Scheduled Visits of the Prehabilitation Prescription Protocol | Up to 18 Weeks
  Feasibility will be measured as the percentage of participants attending scheduled visits of the prehabilitation prescription protocol. Criterion for success: At least (≥) 70% of participants attend all scheduled visits.
Aim 2: Acceptability of Participants That Feel Satisfied with the Prehabilitation Prescription Protocol | Up to 18 Weeks
  Acceptability will be measured as the percentage of participants that report satisfaction with the prehabilitation prescription protocol. Criterion for success: At least (≥) 80% of participants complete the prehabilitation prescription protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Akina Natori, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States